CLINICAL TRIAL: NCT03167619
Title: Phase II Multicenter Study of Durvalumab and Olaparib in Platinum tReated Advanced Triple Negative Breast Cancer
Brief Title: Phase II Multicenter Study of Durvalumab and Olaparib in Platinum tReated Advanced Triple Negative Breast Cancer (DORA)
Acronym: DORA
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Principal Investigator, Sarah Sammons, MD, Assistant Professor of Medicine, Duke University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Pro00080769
Record Dates: First submitted 2017-05-23; First posted 2017-05-30 (Actual); Results first posted 2022-09-13 (Actual); Last update posted 2022-09-13 (Actual); Status verified 2022-06

CONDITIONS: Triple Negative Breast Cancer
Keywords: Metastatic; Platinum Sensitive; Advanced; PARP inhibitor
MeSH Terms: conditions — Triple Negative Breast Neoplasms; Neoplasm Metastasis | interventions — durvalumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- A - olaparib alone (Experimental): Twice daily oral Olaparib 300mg alone as maintenance therapy until disease progression, intolerable toxicity, elective withdrawal from the study, or study completion or termination.
  Interventions: Drug: Olaparib Oral Product
- B - olaparib plus durvalumab (Experimental): Twice daily oral olaparib plus intravenous Durvalumab every 4 weeks as maintenance therapy until disease progression, intolerable toxicity, elective withdrawal from the study, or study completion or termination.
  Interventions: Drug: Olaparib Oral Product in combination with Durvalumab

INTERVENTIONS:
Drug: Olaparib Oral Product — olaparib 300mg twice daily
  Arms: A - olaparib alone
Drug: Olaparib Oral Product in combination with Durvalumab — olaparib 300mg twice daily plus intravenous durvalumab every 28 days
  Arms: B - olaparib plus durvalumab

SUMMARY:
This is a randomized, international, multicenter, Phase II study designed to explore the efficacy of olaparib or olaparib in combination with durvalumab in platinum-treated mTNBC. The primary objectives are to explore olaparib or olaparib in combination with durvalumab as maintenance therapy following clinical benefit with platinum-based therapy in subjects with mTNBC.

DETAILED DESCRIPTION:
Subjects suitable for enrollment into this trial are adult subjects with histologically documented triple negative adenocarcinoma of the breast that is inoperable, locally advanced, or metastatic, and is not amenable to resection with curative intent, and who have received at least 4 cycles of platinum-based chemotherapy in the 1st or 2nd line setting AND derived clinical benefit (CR / PR / SD) per RECIST 1.1 with platinum-based therapy as determined by the treating physician.

Eligible subjects will be randomized to either olaparib or olaparib in combination with durvalumab. Study treatment will continue until disease progression, intolerable toxicity, elective withdrawal from the study, or study completion or termination. Upon treatment discontinuation, subjects will be followed every 2 months for survival.

Although randomization will be used to allocate subjects to either the olaparib or olaparib in combination with durvalumab arm, no comparisons between treatment regimens are planned. The purpose of randomization was to reduce bias due to subject selection into either treatment arm.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 21 years of age
2. ECOG performance status 0-2
3. Inoperable locally advanced or metastatic breast cancer not amenable to resection with curative intent and histologically confirmed to be estrogen receptor (ER) negative, progesterone receptor (PR) negative, and HER2 negative:

   * ER negative status is defined as < 1% tumor cells positive for ER by immunohistochemistry (IHC), irrespective of staining intensity
   * PR negative status is defined as < 1% tumor cells positive for PR by IHC, irrespective of staining intensity

   NOTE: Enrollment is permitted for ER/PR low-expression subjects (defined as ≤ 10%) who are expected to benefit from this trial at the investigator's discretion.
   * HER2 negative status is determined by:
   * IHC 1+, as defined by incomplete membrane staining that is faint/barely perceptible and within > 10% of invasive tumor cells, or
   * IHC 0, as defined by no staining observed or membrane staining that is incomplete and is faint/barely perceptible and within ≤ 10% of the invasive tumor cells, or
   * FISH negative based on:
   * Single-probe average HER2 copy number < 4.0 signals / cell, or
   * Dual-probe HER2/CEP17 ratio < 2.0 with an average HER2 copy number < 4.0 signals / cell
4. Minimum six 1-weekly doses or three 3-weekly doses of platinum chemotherapy (monotherapy or combination therapy at investigator's discretion) with stable disease (SD), partial response (PR) or complete response (CR) to the platinum therapy as assessed by investigator.
5. Has received no more than 2 prior chemotherapy regimens for metastatic breast cancer including current platinum based chemotherapy.
6. Able to provide a representative formalin-fixed, paraffin embedded tumour specimen archival or fresh tissue for correlative studies and biomarker analysis.
7. Hemoglobin ≥ 9.0 g/dL and no blood transfusions in the 28 days prior to study entry. Absolute neutrophil count ≥1,500/mm3. Platelet count ≥100 x 10^9/L.
8. Total bilirubin <1.5 x the upper limit of normal (ULN) with the following exception: subjects with known Gilbert's disease who have serum bilirubin <3 x ULN may be enrolled.
9. Aspartate transaminase (AST) and alanine transaminase (ALT) <2.5 x ULN with the following exceptions: subjects with documented liver or bone metastases may have AST and ALT <5 x ULN.
10. Alkaline phosphatase (ALP) <2 x ULN (<5 x ULN in subjects with known liver involvement and <7 ULN in subjects with known bone involvement).
11. Serum creatinine <1.5 x ULN or creatinine clearance >51 mL/min by the Cockcroft-Gault formula (Cockcroft and Gault 1976) or by 24-hour urine collection for determination of creatinine clearance.
12. For subjects of childbearing potential, agreement (by both subject and partner) to use two effective forms of contraception, including surgical sterilization, reliable barrier method, birth control pills, contraceptive hormone implants, or true abstinence and to continue its use for the duration of the study and for 3 months after last dose of study treatment.
13. Subjects of childbearing potential should have a negative urine or serum pregnancy test during their screening visit. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required.
14. Subjects willing and able to comply with the protocol for the duration of the study including undergoing treatment and scheduled visits and examination.
15. For inclusion in genetic research, subjects must provide informed consent for genetic research collection of specimens to be stored at repository for future research.

Exclusion Criteria:

1. Currently participating and receiving study therapy or has participated in a study of an investigational agent and received study therapy or used an investigation device within 4 weeks of first dose of treatment. Subjects who have entered the follow-up phase of an investigational study may participate as long as it has been 4 weeks since last dose of the previous investigational agent or device.
2. Concurrent enrollment in another clinical study, unless it is an observational (non interventional) clinical study or the follow-up period of an interventional study.
3. Active autoimmune disease that has required systemic treatment in past 2 years (ie, with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (eg, thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, or similar treatment) is not considered a form of systemic treatment.
4. Is taking chronic systemic steroids in doses > 10mg of prednisolone or equivalent within 7 days prior to the first dose of trial treatment.
5. Previous treatment with PARP inhibitors including olaparib.
6. Patients that have required discontinuation of treatment due to treatment-related toxicities from prior therapy with PD-1, PDL-1 or CTLA-4 inhibitors or previous history of immune-related grade 3 or 4 adverse event.
7. Known active central nervous system metastasis and / or carcinomatous meningitis. Subjects with previously treated brain metastases may participate, provided they have:

   1. Stable brain metastases [without evidence of progression by imaging (confirmed by computerized tomography {CT} scan if CT used at prior imaging) for at least four weeks prior to the first dose of trial treatment**,
   2. No evidence of new or enlarging brain metastases; any neurologic symptoms should have returned to baseline,
   3. Not used steroids for brain metastases in the 7 days prior to trial initiation. Taking chronic systemic steroids in doses ≤ 10mg of prednisolone is allowed.

      * This exception does not include carcinomatous meningitis, as subjects with carcinomatous meningitis are excluded regardless of clinical stability.
8. History and/or confirmed pneumonitis, or extensive bilateral lung disease on high resolution/spiral CT scan.
9. Patients with suspected or confirmed myelodysplastic syndrome/acute myeloid leukemia.
10. History of another primary malignancy except for:

    1. Malignancy treated with curative intent and with no known active disease ≥5 years before the first dose of study drug and of low potential risk for recurrence.
    2. Adequately treated non-melanoma skin cancer or lentigo maligna without evidence of disease.
    3. Adequately treated carcinoma in situ without evidence of disease eg, cervical cancer in situ.
11. Major surgery within 2 weeks of starting the study, and subjects must have recovered from any effects of any major surgery.
12. Receipt of radiation therapy within 4 weeks prior to starting study drug(s). Limited field of radiation for palliation within 2 weeks of the first dose of study treatment is allowed provided:

    1. The lung is not in the radiation field
    2. Irradiated lesion(s) cannot be used as target lesions
13. Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, uncontrolled hypertension, unstable angina pectoris, cardiac arrhythmia, active peptic ulcer disease, active bleeding diatheses including any subjects known to have evidence of acute or chronic hepatitis B, hepatitis C or human immunodeficiency virus (HIV), or psychiatric illness / social situations that would limit compliance with study requirements or compromise the ability of the subject to give written informed consent.
14. Subjects unable to swallow orally administered medication, and subjects with gastrointestinal disorders likely to interfere with absorption of the study medication.
15. Subjects requiring treatment with potent inhibitors or inducers of CYP3A4.
16. Pregnant or breast-feeding women. If breastfeeding can be stopped prior to study enrollment until 1 month after the last study dose, then the patient could be allowed to enter the study.
17. Immunodeficient subjects, eg, subjects who are known to be serologically positive for human immunodeficiency virus (HIV).
18. Received a live vaccine within 30 days of planned start of study therapy.
19. Subjects with a known hypersensitivity to olaparib or durvalumab, or any of the excipients of the product.
20. Active or prior documented inflammatory bowel disease (eg, Crohn's disease, ulcerative colitis)
21. History of allogeneic organ transplant
22. Active bleeding diatheses
23. Patients with known active hepatic disease (ie, Hepatitis B or C)
24. Known history of previous clinical diagnosis of tuberculosis.

Min Age: 21 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2018-10-04 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2022-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sarah Sammons, MD, Principal Investigator — Duke Cancer Institute
Locations (1):
- Duke University, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Tan TJ, Sammons S, Im YH, She L, Mundy K, Bigelow R, Traina TA, Anders C, Yeong J, Renzulli E, Kim SB, Dent R. Phase II DORA Study of Olaparib with or without Durvalumab as a Chemotherapy-Free Maintenance Strategy in Platinum-Pretreated Advanced Triple-Negative Breast Cancer. Clin Cancer Res. 2024 Apr 1;30(7):1240-1247. doi: 10.1158/1078-0432.CCR-23-2513. PMID 38236575

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | A - Olaparib Alone | B - Olaparib Plus Durvalumab
Started | 23 | 22
Completed | 11 | 11
Not Completed | 12 | 11
Not completed — Death | 11 | 8
Not completed — Withdrawal by Subject | 1 | 2
Not completed — Physician Decision | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | A - Olaparib Alone | B - Olaparib Plus Durvalumab | Total
Number analyzed (Participants) | 23 | 22 | 45
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.4 (11.9) | 49.5 (11.7) | 51 (11.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23 | 22 | 45
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 22 | 22 | 44
  Unknown or Not Reported | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 16 | 18 | 34
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 5 | 4 | 9
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 2 | 0 | 2

OUTCOME MEASURES:

1. Primary Outcome: Efficacy of Olaparib Alone as Assessed by PFS (Progression-free Survival) Reported as Events Per Month
Description: PFS, defined as the time from randomization to the first occurrence of disease progression or death from any cause on study for olaparib alone. Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1) as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions. Death on study is defined as death from any cause within 30 days of the last dose of study treatment regimen. Reported as events (disease progression or death) per month.
Time Frame: From date of randomization until the date of documented progression or date of death, whichever came first, approximately 1 year.
Population: Intent To Treat population. Only applies to the "olaparib alone" arm.
Measure: Mean (95% Confidence Interval); unit: events/month
Arm/Group | A - Olaparib Alone
Number analyzed (Participants) | 23
events/month | 0.18 [0.11 to 0.27]
Statistical Analysis 1: Comparison: A - Olaparib Alone; Assumed median PFS = 2.0 months as historical control, transformed to rate of 0.35/month; Test type: Superiority; p = 0.0023, Chi-squared; Comparison to mean of historical control; MLE assuming exponential distribution = 0.18, 95% CI 2-sided [0.11 to 0.27] — Presence of patients with long PFS may have violated exponential assumption

2. Primary Outcome: Efficacy of Olaparib in Combination With Durvalumab as Assessed by PFS (Progression-free Survival)
Description: PFS, as defined as the time from randomization to the first occurrence of disease progression (as determined using RECIST v1.1 criteria and assessed by the investigator) or death from any cause on study for olaparib in combination with durvalumab. Death on study is defined as death from any cause within 30 days of the last dose of study treatment regimen. Reported as (disease progression or death) events per month.
Time Frame: as for outcome 1
Population: Intent to Treat population. Only applies to the "olaparib plus durvalumab" arm.
Measure: Mean (95% Confidence Interval); unit: events/month
Arm/Group | B - Olaparib Plus Durvalumab
Number analyzed (Participants) | 22
events/month | 0.11 [0.07 to 0.19]
Statistical Analysis 1: Comparison: B - Olaparib Plus Durvalumab; Assumed median PFS = 2.0 months as historical control, transformed to rate of 0.35/month; Test type: Superiority; p < 0.0001, Chi-squared; Comparison to mean of historical control; MLE assuming exponential distribution = 0.11, 95% CI 2-sided [0.07 to 0.19] — Presence of patients with long PFS may have violated exponential assumption

3. Secondary Outcome: Overall Survival (Olaparib Alone)
Description: To determine the efficacy of maintenance olaparib following platinum based chemotherapy as assessed by overall survival (OS).
Time Frame: From date of randomization until death or last patient contact, approximately 2 years
Population: Only applies to the "olaparib alone" arm.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | A - Olaparib Alone
Number analyzed (Participants) | 23
months | 21.68 [7.69 to NA] — Did not observe enough death events among participants to estimate the upper limit of the 95% CI for median overall survival time.

4. Secondary Outcome: Overall Survival (Olaparib in Combination With Durvalumab)
Description: To determine the efficacy of maintenance olaparib in combination with durvalumab following platinum based chemotherapy as assessed by overall survival (OS).
Time Frame: From date of randomization until death or last patient contact, approximately 2 years
Population: Only applies to the "olaparib plus durvalumab" arm.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | B - Olaparib Plus Durvalumab
Number analyzed (Participants) | 22
months | 18.27 [8.18 to NA] — Did not observe enough death events among participants to estimate the upper limit of the 95% CI for median overall survival time.

5. Secondary Outcome: Overall Response Rate (ORR) as Measured by Number of Participants Achieving Complete Response (CR) or Partial Response (PR) as Defined by RECIST 1.1 (Olaparib Alone)
Description: To determine the efficacy of maintenance olaparib following platinum-based chemotherapy as assessed by overall response rate (ORR) based on RECIST 1.1 (Response Evaluation Criteria In Solid Tumors Criteria). Per RECIST v1.1 for target lesions and assessed by CT or MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR.
Time Frame: Assessed every 8 weeks from date of randomization until documented disease progression or last patient contact, approximately 1 year
Population: Only applies to the "olaparib alone" arm.
Measure: Count of Participants; unit: Participants
Arm/Group | A - Olaparib Alone
Number analyzed (Participants) | 23
Participants | 5

6. Secondary Outcome: Overall Response Rate (ORR) as Measured by Number of Participants Achieving Complete Response (CR) or Partial Response (PR) as Defined by RECIST 1.1 (Olaparib in Combination With Durvalumab)
Description: To determine the efficacy of maintenance olaparib in combination with durvalumab following platinum-based chemotherapy as assessed by overall response rate (ORR) based on RECIST 1.1 (Response Evaluation Criteria In Solid Tumors Criteria). Per RECIST v1.1 for target lesions and assessed by CT or MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR.
Time Frame: as for outcome 5
Population: Only applies to the "olaparib plus durvalumab" arm.
Measure: Count of Participants; unit: Participants
Arm/Group | B - Olaparib Plus Durvalumab
Number analyzed (Participants) | 22
Participants | 3

7. Secondary Outcome: Clinical Benefit Rate (CBR) as Measured by the Number of Participants Achieving Complete Response (CR), Partial Response (PR) or Stable Disease for ≥ 24 Weeks (SD) as Defined by RECIST 1.1. (Olaparib Alone)
Description: To determine the efficacy of maintenance olaparib following platinum-based chemotherapy as assessed by clinical benefit rate (CBR) based on RECIST 1.1 (Response Evaluation Criteria In Solid Tumors Criteria). Per RECIST v1.1 for target lesions and assessed by CT or MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Stable Disease (SD), neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for Progressive Disease (PD); Clinical Benefit (CB) = CR + PR + SD for >= 24 weeks.
Time Frame: as for outcome 5
Population: Only applies to the "olaparib alone" arm.
Measure: Count of Participants; unit: Participants
Arm/Group | A - Olaparib Alone
Number analyzed (Participants) | 23
Participants | 9

8. Secondary Outcome: Clinical Benefit Rate (CBR) as Measured by the Number of Participants Achieving Complete Response (CR), Partial Response (PR) or Stable Disease for ≥ 24 Weeks (SD) as Defined by RECIST 1.1. (Olaparib in Combination With Durvalumab)
Description: To determine the efficacy of maintenance olaparib in combination with durvalumab following platinum-based chemotherapy as assessed by clinical benefit rate (CBR) based on RECIST 1.1 (Response Evaluation Criteria In Solid Tumors Criteria). Per RECIST v1.1 for target lesions and assessed by CT or MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Stable Disease (SD), neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for Progressive Disease (PD); Clinical Benefit (CB) = CR + PR + SD for >= 24 weeks.
Time Frame: as for outcome 5
Population: Only applies to the "olaparib plus durvalumab" arm.
Measure: Count of Participants; unit: Participants
Arm/Group | B - Olaparib Plus Durvalumab
Number analyzed (Participants) | 22
Participants | 8

ADVERSE EVENTS:
Time Frame: From the first dose of either study drug through 30 days after the last dose of either study drug or until the initiation of an alternative anticancer therapy, up to 2 years
Arm/Group | A - Olaparib Alone | B - Olaparib Plus Durvalumab
All-Cause Mortality (participants affected / at risk) | 11/23 | 8/22
Serious Adverse Events (participants affected / at risk) | 2/23 | 3/22
Other Adverse Events (participants affected / at risk) | 23/23 | 21/22
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | A - Olaparib Alone (N=23) | B - Olaparib Plus Durvalumab (N=22)
Pyrexia (General disorders) | 0 | 2
Nausea (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 1
Pneumonia (Infections and infestations) | 0 | 1
Neutrophil count decreased (Investigations) | 0 | 1
Tumour associated fever (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | A - Olaparib Alone (N=23) | B - Olaparib Plus Durvalumab (N=22)
Nausea (Gastrointestinal disorders) | 13 | 9
Fatigue (General disorders) | 12 | 6
Anaemia (Blood and lymphatic system disorders) | 9 | 7
Decreased appetite (Metabolism and nutrition disorders) | 6 | 9
Vomiting (Gastrointestinal disorders) | 5 | 7
Dizziness (Nervous system disorders) | 6 | 5
Diarrhoea (Gastrointestinal disorders) | 4 | 5
Neutrophil count decreased (Investigations) | 5 | 4
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 7
Headache (Nervous system disorders) | 2 | 6
Mucosal inflammation (General disorders) | 4 | 3
Constipation (Gastrointestinal disorders) | 4 | 2
Peripheral sensory neuropathy (Nervous system disorders) | 2 | 4
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 | 3
Platelet count decreased (Investigations) | 2 | 3
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 3
Insomnia (Psychiatric disorders) | 3 | 2
Rash (Skin and subcutaneous tissue disorders) | 3 | 2
Pain (General disorders) | 2 | 2
Pyrexia (General disorders) | 1 | 3
White blood cell count decreased (Investigations) | 2 | 2
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 | 3
Neutropenia (Blood and lymphatic system disorders) | 2 | 1
Dry mouth (Gastrointestinal disorders) | 0 | 3
Dyspepsia (Gastrointestinal disorders) | 2 | 1
Influenza like illness (General disorders) | 1 | 2
Non-cardiac chest pain (General disorders) | 1 | 2
Pneumonia (Infections and infestations) | 2 | 1
Blood creatinine increased (Investigations) | 3 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 2
Hypothyroidism (Endocrine disorders) | 0 | 2
Oral pain (Gastrointestinal disorders) | 0 | 2
Chills (General disorders) | 0 | 2
Alanine aminotransferase increased (Investigations) | 2 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 2 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Hypertension (Vascular disorders) | 2 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-06-14): https://cdn.clinicaltrials.gov/large-docs/19/NCT03167619/Prot_SAP_000.pdf